CLINICAL TRIAL: NCT00688337
Title: Correlation Between Fluorodeoxyglucose (FDG) and FLT Uptake and Gene-Expression Oncotype Assay in Patients With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Einat Even-Sapir MD, PhD, Dept of Nuclear Medicine, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-08-EE-108-CTIL
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; lymph nodes; gene-expression; oncotype; Age over 18; Newly diagnosed breast cancer prior to surgery or treatment.; No evidence of clinical nodal disease
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — not relevant
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients with newly diagnosed breast cancer. Clinically nodal negative.

SUMMARY:
In the current study FDG (Fluorodeoxyglucose) uptake, FLT uptake (F18-Fluoro-3'-deoxythymidine) and their ratios will be correlated with the risk score results of the Oncotype gene-expression assay in patients with clinically negative nodal disease planned for surgical removal of the tumor.

DETAILED DESCRIPTION:
Several publications have addressed the role of PET imaging for biological characterization of breast cancer. A modest but significant correlation was reported between tumor grading and FDG uptake. Few studies reported a positive correlation between SUV and the Ki-67 labeling index of malignant breast tumors. Others have correlated p53 expression in breast cancer and FDG uptake. F18-Fluoro-3'-deoxythymidine (FLT) has been developed as a PET marker for cellular proliferation has been developed for imaging cell proliferation and findings correlate strongly with the Ki-67 labeling index in breast cancer. A 10-minute FLT-PET scan acquired two weeks after the end of the first course of chemotherapy, has been shown in two recent studies to be useful for predicting longer-term efficacy of chemotherapy regimens for women with breast cancer.

In the current study FDG and FLT uptake and their ratios will be correlated with the risk score results of the Oncotype gene-expression assay in patients with clinically negative nodal disease planned for surgical removal of the tumor. It is our hypothesis that since high uptake of these tracers implies aggressive behavior and rapid tumor growth, it might well be that patients with high risk score on Oncotype will have high uptake of the PET tracers and those with low risk score will show low-intensity uptake values. If this will be the case, it might well be that in patients with non-conclusive oncotype results (intermediate score) FDG and FLT uptake measurement will allow further dichotomy to 1. Patients with intermediate score on Oncotype and high uptake of the PET tracers, suggestive of aggressive behavior and 2. Patients with intermediate score on Oncotype and low uptake of the PET tracers suggesting a less aggressive behavior.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with breast cancer
* clinically nodal negative
* prior to surgery and/or treatment
* age over 18 years

Exclusion Criteria:

* Age under 18
* Pregnancy
* Previous therapy for breast cancer
* Clinical or histological evidence of nodal involvement or other proven metastatic sites

Ages: 18 Years to 86 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients with breast cancer, clinically nodal negative, prior to surgery and/or treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between FDG and FLT uptake and hystological findings and Oncotype results | One year after imaging

SECONDARY OUTCOMES:
Clinical outcome | A year after imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel